CLINICAL TRIAL: NCT05853653
Title: The Effect of Breastfeeding Education Using a Doll During Pregnancy on Newborn Feeding: A Randomized Control Trial
Brief Title: The Effect of Breastfeeding Education Using a Doll During Pregnancy on Newborn Feeding
Acronym: Newborn
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Istinye University (Other)
Responsible Party: Principal Investigator, Aysegul Simsek, Assist. Prof. Dr., Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IstinyeU; NCT06197633 (obsolete NCT alias)
Record Dates: First submitted 2023-04-04; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Breastfeeding Education; Newborn; Vitality; Education
Keywords: Breastfeeding; Nutrition; Newborn; Breastfeeding education; Education with a material
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Randomized controlled quasi-experimental design
Who Masked: Participant
Masking Description: Single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Using dolls in breastfeeding education (Experimental): In the breastfeeding training, the researchers will explain the pre-created training content. It will then be demonstrated practically using the baby. A training brochure will be given at the end of the training.
  Interventions: Behavioral: Using dolls in breastfeeding education
- Verbal expression is used in breastfeeding education (No Intervention): In the breastfeeding training, the researchers will verbally explain the pre-created training content. A training brochure will be given at the end of the training.

INTERVENTIONS:
Behavioral: Using dolls in breastfeeding education — Using dolls in breastfeeding education
  Arms: Using dolls in breastfeeding education

SUMMARY:
This study was planned in a randomized controlled quasi-experimental design to determine the effect of breastfeeding education using a doll during pregnancy on newborn feeding. Necessary institutional and ethics committee permissions will be obtained before the study. Before data collection, the consent form will be read to the pregnant women who meet the inclusion criteria and volunteer to participate in the study and their written and verbal consent will be obtained. The information in the participant information form will be questioned before the training. In the prenatal period of the study, the Control group will be given the standard breastfeeding education applied by the institution verbally. In the intervention group, breastfeeding education prepared in line with the relevant literature will be given by the researchers. Individual breastfeeding training will be given to each participant by a researcher.

DETAILED DESCRIPTION:
The most important nutrient in infant nutrition has been breast milk throughout history. Breastfeeding has many benefits for both the infant, the mother and the society. In addition to reducing mortality and morbidity rates in infants, it provides a healthy growth and development process. It has positive effects on the mother such as feeling happy, being physically healthy with the effect of hormones, facilitating the return of the uterus, providing emotional satisfaction, reducing the risk of breast cancer, reducing the risk of anemia, reducing the risk of depression, facilitating mother-infant bonding, and protecting from a new pregnancy. In addition, being free and natural, decreasing maternal-infant mortality, decreasing the risk of disease, providing healthy individuals to the society, being fast and requiring preparation, decreasing health expenditures, decreasing the loss of labor force, decreasing the risk of loss of money for working mothers were the benefits to the society and the country. In the world and in our country, many practices are carried out to popularize breastfeeding. One of the most important of these practices is the friendly hospital practice, which informs pregnant women and families about the importance of breastfeeding. Skin-to-skin contact between mother and baby is ensured immediately after birth, and the mother is supported to start breastfeeding as soon as possible and not to interrupt contact (Bolat et al, 2011; Samur, 2006). This approach aims to increase the rate of breastfeeding. However, in the changing world order, there may be problems in maintaining the maternal herd due to the inclusion of women in business life. For this reason, practices to promote breastfeeding are on the agenda. The primary aim of these practices is to provide exclusive breastfeeding for the first 6 months, supplementary feeding from the 6th month onwards and continuation of breastfeeding until the age of 2 years. Within the scope of the "Promotion of Breastfeeding and Baby Friendly Hospitals Program" in our country, it is aimed to reach all hospitals where births are performed and to provide education and information in these hospitals. For this reason, prenatal and postnatal breastfeeding and breastfeeding education is provided by health professionals. It is also recommended that this education should be shaped according to the needs of women, the content should be diversified, teaching should be carried out by using technology, and continuity of education should be ensured.

ELIGIBILITY:
Inclusion Criteria:

* Being in the last trimester of pregnancy
* Having a healthy pregnancy
* Fetus and newborn are healthy
* Having the mother and baby in the same room in the postpartum period

Exclusion Criteria:

* Not knowing Turkish
* The woman has neurological and cognitive problems
* Hearing and vision problems in the woman

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 209 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Effective use of dolls and breastfeeding education | 6 months
  The effect of breastfeeding education using dolls will be obtained by analyzing the data collected with data collection tools.
Effect of breastfeeding education on breastfeeding self-efficacy level | 6 months
  The effect of breastfeeding education on the level of breastfeeding self-efficacy will be obtained by analyzing the data.

CONTACTS AND LOCATIONS:
Overall Officials: Aysegul Simsek, PhD, Principal Investigator — Istinye University
Locations (1):
- Aysegul Simsek, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
It can be shared with a reasonable request from the principal investigator after the study is published.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after the study is published in a journal.
Access Criteria: A reasonable request

REFERENCES:
- [Background] Arça G, Işık HK (2019) The role of midwife and nurse regarding breast milk and breastfeeding Health Sciences University Nursing, 2019;3(1): 221-228.
- [Background] Eksioglu AB, Ceber E. Translation and validation of the Breast-feeding Self-efficacy Scale into Turkish. Midwifery. 2011 Dec;27(6):e246-53. doi: 10.1016/j.midw.2010.10.009. Epub 2010 Dec 8. PMID 21145148
- [Background] Bolat F, Uslu S, Bolat G, Bülbül A, Arslan S, Çelik M, Cömert S, Nuhoğlu A (2011) Factors affecting breastfeeding in the first six months. Çocuk Dergisi, 11(1):5-13. doi:10.5222/j.child.2011.005
- [Background] Samur G. Nutrition in Pregnancy and Lactation. T.C. Ministry of Health, General Directorate of Primary Health Care Services, Department of Food Safety, Nutrition Information Series. 2006, 1st Edition. Sinem Matbaacılık, Ankara
- [Background] Yılmaz M, Kaya NY, Çiçek H, Şahin H, İnanç N, Akyut M (2012) The Effect of Breastfeeding Education Given During Pregnancy on Breastfeeding and Breastfeeding Related Behaviors. Journal of Nutrition and Diet 2012;40(1):2-11